CLINICAL TRIAL: NCT05943951
Title: Lymphadenectomy in Right Hemicolectomy: Italian Multicenter Study (CoDIG-2)
Brief Title: Italian Study on the Right Hemicolectomy: How the Lymphadenectomy is Performed
Acronym: CoDIG-2
Status: Completed | Type: Observational
Sponsor: Gabriele Anania (Other)
Responsible Party: Sponsor-Investigator, Gabriele Anania, Prof., University Hospital of Ferrara
Organization: University Hospital of Ferrara (Other)
Other Study IDs: CoDIG-2
Record Dates: First submitted 2023-06-27; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Colon Cancer; Lymph Node Metastasis; Surgical Procedure, Unspecified
Keywords: Right hemicolectomy; Colon cancer; Lymphadenectomy
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Right hemicolectomy — It begins with a thorough laparoscopic inspection of the abdomen for evidence of metastatic disease and to confirm the location of the tumor. Usually is performed dissection using a medial-to-lateral approach. A lateral or inferior approach can also be used depending on the anatomy. The vascular dissection may begin at the ileocolic pedicle or over the superiore mesenteric vein. After completing the medial-to-lateral dissection, the sourgeons return to the ileocolic pedicle to begin vascular dissection. Whether a D2 (until encountering the right branch of the middle colic) or D3 dissection (until the root of ileocolic artery and vein) is performed depends upon the tumor stage. For an intracorporeal anastomosis, the bowel is transected proximally and distally using a linear stapler. The terminal ileum is positioned along the transverse colon in an isoperistaltic fashion. After that a colotomy and an enterotomy are made on the antimesenteric edge of the colon and small bowel respectively

SUMMARY:
The objective of the study is the analysis of lymphadenectomy in the course of right hemicolectomy, in relation to the radicality of the surgical resection that is performed. In particular, the investigators wants to inquire how according to precise standards regarding surgical radicalness and consequently the anatomical piece that is obtained it is possible to correlate a certain number of lymph nodes and their possible positivity.

The lead center is the General and Thoracic Surgery Department of the University of Ferrara. Prof. Anania is the responsible for the enrollment of patients and the coordination with the collaborating centers in the six month-study

DETAILED DESCRIPTION:
All the high-volume specialist centres that perform this type of intervention in Italy will be invited, with a minimum number of 25 interventions per year. At the end of the study 788 patients was enrolled.

The data of the patients involved will be collected independently and anonymously by the individual centers involved, using a common alpha numeric code decided by the coordinating center.

The parameters examined will be:

* Personal data of the patient
* Stage of neoplasm due to surgery
* Type of surgery and duration
* Post-operative course
* Presence of post-surgical complications and eventual hospital readmission due to these complications
* Study of the operating piece and lymphadenectomy performed:

Tumor free margin Terminal ilium length The different vascular ligatures and levels at which they are performed Integrity of the mesocolon Number of positive nodes per total removed

Following the end of the 6 months of observational study period, the data will be processed anonymously at the coordinating centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients and/or legal guardians, where applicable, have been fully informed and have voluntarily provided informed written consent or patients unable to read and/or write who have fully understood the information verbally provided by the investigator and who have provided a verbal consent testified in writing by a third person.

  * Patients aged > 18, men and women, operated by laparoscopic right hemiolectomy or video assisted, under election regime at the U.O. General and Thoracic Surgery with diagnosis of colic adenocarcinoma at any stage.
  * Patients who have already undergone chemotherapy and radiotherapy for other reasons.

Exclusion Criteria:

* Under age.
* Patients undergoing emergency surgery.
* Women who are pregnant.
* Patients with right-handed laparotomy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18, men and women, operated by laparoscopic/robotic or video-assisted right hemicolectomy, under election regime with diagnosis of colic adenocarcinoma in one of the centers that take part of the study After the 6 months period a total of 788 patients was enrolled in the 76 italian centers
Sampling Method: Non-Probability Sample
Enrollment: 788 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
the analysis of lymphadenectomy in the course of right hemciolectomy, in relation to the radicality of surgical resection that is performed | 6 months
  In particular, the invastigators want to inquire how according to precise standards regarding surgical radicalness and consequently the anatomical piece that is obtained it is possible to correlate a certain number of lymph nodes and their possible positivity. In the study various items about lymphadenectomy will be invastigated: tumor free margin > 5cm, lenght of teminal ileum > 10cm, different level at which colic vessel are closed (proximal or distal ligation) and consequentially the different lymph nodes stations collected, mesocolic sail integrity based on Benz score, number of lymph node harvest and number of lymph nodes positive for metastatic involvement, type of surgical procedure (video-assisted, laparoscopic, robotic).

SECONDARY OUTCOMES:
Vascular anatomical variability | 6 months
  The investigators wants to study the vascular anatomical variability of the patients enrolled in the study, and how this variability may affect the extent of lymphoadenectomy. The investigators will analize the vessels anatomy with pre-operative imaging (CT scan) and with intra-operative feedback. The attention will be on the position of superior mesenteric artery relative to superior mesenteric vein (before or behind). Futhermore the invastigators wants to study the anatomical variants of the vessels: the presence of the middle colic artery and its branches, the presence of the right colic artery and their variability in percentage terms

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Anania, Principal Investigator — Ferrara University Hospital
Locations (62):
- Italy (62):
  - Ospedale Carlo Urbani, Iesi, Ancona
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti, Bari
  - IRCCS Saverio de Bellis, Castellana Grotte, Bari
  - Policlinico San Marco Zingonia, Osio Sotto, Bergamo
  - Ospedale Valcamonica, Esine, Brescia
  - ASST Spedali Civili, Montichiari, Brescia
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Firenze
  - Ospedale Nuovo di Legnano, Legnano, Milano
  - Ospedale San Giovanni di Dio Frattamaggiore, Frattamaggiore, Napoli
  - Ospedale Immacolata Concezione Piove di Sacco ULSS 6, Piove di Sacco, Padova
  - Ospedale San Paolo, Civitavecchia, Roma
  - Ospedale CTO, Iglesias, Sud Sardegna
  - Ospedale San Valentino, Montebelluna, Treviso
  - Ospedale di Latisana, Latisana, Udine
  - Ospedale San Pietro e Paolo, Borgosesia, Vercelli
  - Ospedale Umberto I, Ancona
  - Ospedale Bonomo, Andria
  - Ospedale Regionale U. Parini, Aosta
  - Policlinico Ponte San Pietro, Bergamo
  - ASL Biella, Biella
  - IRCCS AOU Bologna, Sant'Orsola, Bologna
  - Ospedale centrale di Bolzano, Bolzano
  - Azienda Ospedaliero universitaria di Cagliari, Cagliari
  - PO Santissima Trinità ASL Cagliari, Cagliari
  - AOU Mater Domini Università Magna Grecia Catanzaro, Catanzaro
  - Anania Gabriele, Ferrara
  - AOU Careggi, Florence
  - Ospedale San Giovanni di Dio, Florence
  - Azienda Ospedaliero Universitaria di Foggia, Foggia
  - Ospedale Morgagni-Pierantoni, Forlì
  - P.O. San Salvatore, L’Aquila
  - Ospedale civile di Macerata, Macerata
  - AO Papardo, Messina
  - IRCCS Ca Granada Ospedale Maggiore Policlinico Milano, Milan
  - Ospedale San Raffaele, Milan
  - AOU Modena, Modena
  - AORN dei Colli - Ospedale Monaldi, Napoli
  - AOU Federico II di Napoli, Napoli
  - Isitituto Nazionale Tumori ICRSS Fondazione G. Pascale, Napoli
  - Policlinico P. Giaccone, Palermo
  - Ospedali Riuniti Marche Nord, Pesaro
  - Ospedale Civile Santo Spirito, Pescara
  - Azienda Ospedaliero Universitaria di Pisa, Pisa
  - Ospedale Santo Stefano, Prato
  - AOU Tor Vergata, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Ospedale San Carlo di Nancy, Roma
  - Ospedale San Filippo Neri ASL Roma 1, Roma
  - Ospedale Sandro Pertini, Roma
  - Ospedale Sant'Andrea, Roma
  - Policlinico Campus biomedico, Roma
  - Ospedale Santa Maria della Misericordia, Rovigo
  - Azienda Ospedaliero Universitaria Sassari, Sassari
  - Ospedale San Paolo, Savona
  - Ospedale Maria Vittoria, Torino
  - Ospedale Martini, Torino
  - Piccola casa della divina provenienza Ospedale Cottolengo, Torino
  - Ospedale Sant'Antonio Abate, Trapani
  - Ospedale San Camillo, Trento
  - AOU Trieste, Trieste
  - Ospedale Sant'andrea, Vercelli
  - Ospedale Belcolle, Viterbo

IPD SHARING:
Plan to Share IPD: No
privacy

REFERENCES:
- [Derived] Anania G, Chiozza M, Campagnaro A, Bagolini F, Resta G, Azzolina D, Silecchia G, Cirocchi R, Agrusa A, Cuccurullo D, Guerrieri M; SICE CoDIG (ColonDx Italian Group). Laparoscopic right hemicolectomy: a SICE (Societa Italiana di Chirurgia Endoscopica e Nuove tecnologie) network prospective study on the approach to right colon lymphadenectomy in Italy: is there a standard?-CoDIG 2 (ColonDx Italian Group). Surg Endosc. 2024 Mar;38(3):1432-1441. doi: 10.1007/s00464-023-10607-8. Epub 2024 Jan 8. PMID 38191814